CLINICAL TRIAL: NCT02501369
Title: A Case Series Examining the Impact of a Positive Parenting Program (Self Directed Teen Triple P) on Treatment Adherence in Families With an Adolescent With Cystic Fibrosis
Brief Title: Investigating the Use of a Positive Parenting Programme to Improve Treatment Adherence in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emma Wells (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor-Investigator, Emma Wells, Trainee Clinical Psychologist, University of Manchester
Organization: University of Manchester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15059
Record Dates: First submitted 2015-05-08; First posted 2015-07-17 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Self-directed Teen Triple P (Experimental): Self-directed Teen Triple P is a behaviourally based parenting intervention that parents follow at home using a workbook. It is based upon social learning theory principles and is used to help parents build upon their existing skills and information to practice positive parenting. Key skills promoted include: Increasing positive parent-teenager interactions, increase desirable behaviour, teach new behaviours and skills, and manage problem behaviour.
  As this is a case series design participants will act as their own controls and so there are no other arms to the study.
  Interventions: Behavioral: Self-directed Teen Triple P

INTERVENTIONS:
Behavioral: Self-directed Teen Triple P — Manualised parenting programme that parents will complete at home. This involves reading weekly modules of the manual and completing small exercises to practice the skills taught. These include strategies to help build positive relationships between parent and child, helping parents to effectively manage challenging childhood behaviours, and providing parents with the skills to support their child's independence and independent management of their cystic fibrosis.

SUMMARY:
Cystic fibrosis (CF) is an illness that makes the lungs clog up with sticky mucus. There is no cure and so treatments are used to help make the illness easier to live with. The treatment can take lots of time and can feel not very nice sometimes. When children with CF become teenagers they need to learn to take charge of their treatment. This can be difficult. Teenagers with CF want to fit in with friends and can become more upset about their illness. Their parents have to learn to let their child take charge of their illness which can be hard for parents. These issues can put strain on parent-child relationships and this can make it harder for teenagers to stick to their treatment plans. A parenting program (called Teen Triple P) has been shown to help teenagers with other illnesses (such as diabetes) to be able to stick to their treatment plans. Parents are given a booklet to work through at home which helps them to build on the skills they already have. It aims to help families to support positive parent-child relationships, to manage difficult teenage behaviours, and to teach new skills and behaviours. So far no one has done any research to see if this program helps families of teenagers with CF. This research would like to see if the Triple P program can help teenagers with CF stick to their treatment plan. Helping teenagers stick to their treatment plan will help them to live happier and healthier lives.

DETAILED DESCRIPTION:
The aim of this case series is to begin to explore whether the Teen Triple P program may improve treatment adherence, parent-child relationships, parenting experiences and parent and adolescent wellbeing in families with an adolescent with CF. Research commonly reports that adherence rates to treatment are consistently lower in this age group, with variables such as parent-child conflict, parent stress and the child's increasing independence all being influential factors. Previous research has suggested that family based interventions may facilitate with treatment adherence in this population, but little research has investigated the effectiveness of specific parenting and family based interventions. Triple P is an internationally recognized and extensively researched parenting intervention that has been found to support families from an array of clinical and non-clinical samples, and has been shown to reduce family conflict in other chronic health conditions. No research to date has examined the use Triple P interventions in cystic fibrosis and so hence the current research.

A within subjects clinical case series using an A-B multiple baseline design will be used. This type of design exposes participating parents to a multiple baseline period (phase A) followed by an intervention phase (phase B). This controls for potential confounds, which increases confidence that change is attributable to the use of the parenting intervention. The baseline phase will vary in length from 2 to 6 weeks. During this phase, parents will complete the treatment adherence questionnaire and parenting scale (outlined in the outcome measures section) at weekly intervals which will take 10 minutes each week (the first and last baseline session will involve completing all questionnaires stated in the primary and secondary outcome measures section). The baseline phase will be followed by the 10 week intervention phase. Here parents will commence the self-directed Teen Triple P programme. Parents will be posted a copy of the Teen Triple P workbook. They will complete a 1 hour module of Triple P each week and will also continue to complete the treatment adherence questionnaire and parenting scale each week. At week 5 and 10 of the intervention, the full set of outcome questionnaires will be administered, as well as a satisfaction survey to determine how parents are finding the Triple P intervention. Once the 10 week Triple P intervention has been completed a period of 4 weeks will elapse before the researcher will contact the parents again in order for them to complete a set of 1 month follow up questionnaires, as well as answering some questions about their experiences of taking part in the Triple P intervention.

Children themselves will not be required to participate in any study related activity as this is primarily a parenting intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parents of adolescents (aged 11 to 16) with Cystic Fibrosis.
* Self reported difficulties with their child's treatment adherence.

Exclusion Criteria:

* Families already receiving psychological support from specialist Cystic Fibrosis clinical psychologists
* Parents requiring reading assistance who do not have anyone to help them
* Families where the parent/ child is currently being treated for a mental health difficulty

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Treatment Adherence from baseline as measured by Treatment Adherence Questionnaire - Revised (Quittner et al., 2008) | baseline, intervention weeks 1, 2,3,4,5,6,7,8,9,10, and 1 month follow up
  consists of 12 items across four subscales corresponding to different domains of CF treatment regime. It asks about adherence to various elements of treatment in the last week. Answers are measured across a 6 point Likert scale ranging from "not at all" to "3 or more times a day". Internal consistency (α=.82-.84) and test-retest reliability (r's=.42-.57) have been examined. This measure takes a maximum of 5 minutes to complete.
Change in parenting skill and competence from baseline as measured by The Parenting Scale (PS; Arnold et al., 1993) | baseline, intervention weeks 1, 2,3,4,5,6,7,8,9,10, and 1 month follow up
  30 item questionnaire measuring parent discipline styles. It has adequate internal consistency, good test-retest reliability and reliably distinguishes between clinical and non-clinical samples. This measure takes approximately 10 minutes to complete.

SECONDARY OUTCOMES:
Change in parent stress from baseline as measured by Pediatric Inventory for Parents: PIP (Streisand et al., 2001) | baseline,weeks 5 and 10 of intervention, and 1 month follow-up
  This has 42 items that ask parents to describe the frequency and intensity with which they experience stress related to caring for their child's illness across four domains: (a) communication (b) emotional functioning (c) child's medical care and (d) role functioning. Parents indicate on a scale from 1 (never) to 5 (very often) how often an event had occurred in the past 7 days and how difficult each event was. Internal consistency for the PIP has been shown to be good for both scales, frequency: α = .94, difficulty: α = .96
Change in parent's sense of competence from baseline as measured by Parent Sense of Competency Scale (PSOC; Gibaud-Wallston & Wandersman, 1978) | baseline,weeks 5 and 10 of intervention, and 1 month follow-up
  A 17 item measure assessing parental competence on two dimensions: satisfaction with the parenting role and feelings of efficacy as a parent. This also has good internal consistency and test-retest reliability. This measure takes approximately 5 minutes to complete
Change in child's emotional wellbeing and behavioural difficulties from baseline as measured by Strengths and Difficulties Questionnaire (SDQ: Goodman, 1997) | baseline,weeks 5 and 10 of intervention, and 1 month follow-up
  a brief behavioural screening questionnaire about 3-16 year olds. Parents are asked 25 questions about their child, which are divided between 5 subscales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behaviour. Parents rate each item as "not true", "somewhat true", and "always true" of their child. This measure has very good psychometric properties and is used as a routine child wellbeing outcome measure in many child mental health teams in the UK.
Change in parent emotional wellbeing from baseline as measured by The Depression, Anxiety and Stress Scale - 21 item version (DASS-21) | baseline,weeks 5 and 10 of intervention, and 1 month follow-up
  a 21 item self-report Questionnaire designed to measure the severity of a range of symptoms common to both Depression and Anxiety. Parents rate their responses to each item on a 4 point Likert scale from "never" to "almost always". The reliability and validity of this measure is very good, with internal consistency and validity being scored in the acceptable to excellent ranges

OTHER OUTCOMES:
Parent satisfaction with the intervention at mid and end intervention points as measured by Client Satisfaction Questionnaire | weeks 5 and 10 of intervention
  is designed to collect information to evaluate the different interventions and help to improve the Triple P programme. Administered only at post-intervention the questionnaire addresses the quality of the intervention, the extent to which it met the participant's needs, the effect it had on their parenting skills and child's behaviour problems. All items are measured on a 7 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Calam, PhD, Principal Investigator — University of Manchester